CLINICAL TRIAL: NCT04732624
Title: Implementation of an Enteral Resuscitation Bundle for Moderate-sized Burn Injuries (20-40% Total Body Surface Area) to Prevent Shock, Coagulopathy, and Kidney and Lung Injury in Nepal
Brief Title: Enteral Resuscitation Nepal (Pilot Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Kajal Mehta, MD MPH, Global Health Research Fellow, School of Medicine: Surgery, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010934; D43TW009345 (NIH)
Record Dates: First submitted 2021-01-20; First posted 2021-02-01 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Burn Body Region Unspecified; Burn Shock
Keywords: Burns; Enteral Resuscitation; Oral Rehydration Solution; Burn Shock; Austere Conditions; Low- and middle-income country
MeSH Terms: conditions — Burns; Osteoarthritis | interventions — World Health Organization oral rehydration solution; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Feasibility study of randomized trial of enteral-based resuscitation (intervention arm) vs. IV fluid resuscitation (standard-of-care arm) for moderate sized burn injuries.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enteral-based Protocolized Resuscitation (Experimental): Administration of Enteral-based Resuscitation using Oral Rehydration Solution (ORS) either by mouth of via naso-enteric access for moderate sized burn injuries (20-40% TBSA) per resuscitation protocol for burn-injured patients. Resuscitation will be administered in the acute resuscitation phase of burn injury (24-72 hours post injury). Patients will receive supplemental Intravenous Fluid (IV Fluid) resuscitation using Lactated Ringer's solution as needed per protocol.
  Interventions: Drug: Oral Rehydration Solution; Drug: Lactated Ringer
- Intravenous Fluid Protocolized Resuscitation (Active Comparator): Administration of Intravenous Fluid using Lactated Ringer's solution per standard of care resuscitation protocol for patients with moderate sized burn injuries (20-40% TBSA).
  Interventions: Drug: Lactated Ringer

INTERVENTIONS:
Drug: Oral Rehydration Solution — Feasibility study of Enteral-based resuscitation with Oral Rehydration Solution (ORS) vs standard-of-care Intravenous Fluid resuscitation for moderate-sized burn injuries in Nepal
  Other Names: Enteral-based Resuscitation
  Arms: Enteral-based Protocolized Resuscitation
Drug: Lactated Ringer — Standard-of-care Intravenous Fluid resuscitation
  Other Names: Intravenous Fluid Resuscitation

SUMMARY:
Nepal and the South Asian sub-continent carry some of the highest rates of burn injury globally, with an associated high morbidity and mortality. Nepal currently has one major center equipped for burn care, in Kirtipur, Nepal and receives referred patients from around the country. At presentation, most patients with major burns have had minimal to no resuscitation on arrival, often hours to days after the burn injury was sustained.

Timely fluid resuscitation, initiated as soon as possible after major burn injury, is the main tenet of acute burn care. Lack of adequate resuscitation in major burn injuries leads to kidney injury, progression of burn injury, sepsis, burn shock, and death. The current standard of care for major burn resuscitation is intravenous fluid resuscitation. In Nepal, however, adequately trained and equipped hospitals for treatment of burn care are not available (for a variety of reasons). Additionally, there is not a systematic emergency medical transport system available for provision of medical care and resuscitation during transport. Enteral-based resuscitation with substances like the WHO Oral Rehydration Solution (ORS) is recommended by burn experts and the professional burn societies when resources and access to intravenous fluid resuscitation are not available in resource-constrained settings such as rural areas, low- and middle-income countries, and military battlefield scenarios. Studies have previously demonstrated the efficacy and safety of enteral-based resuscitation in controlled, high-resource settings, however there have not been real-world effectiveness trials in austere settings. Therefore, the investigators seek to ultimately address the problem of pre-hospital and pre-burn center admission resuscitation by studying the feasibility and effectiveness of enteral resuscitation with Oral Rehydration Solution (ORS) in preventing burn shock.

This study examines enteral (oral)-based resuscitation with ORS and IV Fluids versus only IV Fluids for the treatment of major burn injuries. The intervention portion of the study will entail randomization of patients presenting with acute burn injuries of 20-40% total body surface area (TBSA) to an enteral-based resuscitation versus the standard of care IV fluid resuscitation. The intervention will continue through the 24-72 hours of the acute resuscitation period.

This is a feasibility study, primarily to develop and establish the research infrastructure and practices at the study site for future pilot study and eventually randomized-controlled trial research on this intervention. The primary outcomes will be measures of feasibility such as the adherence rate to the resuscitation protocols. Further, there will be a qualitative component to the study with focus group interviews of the bedside healthcare providers (doctors and nurses) who are caring for the enrolled patients, in order to understand the challenges and facilitators of enteral resuscitation. Qualitative analysis will be done to understand the major themes of challenges and facilitators to enteral resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* All genders
* Adults aged ≥18 years who present with moderate-sized burn injuries [20 - 40% total body surface areas (TBSA)] to the Nepal Cleft and Burn Center within 24 hours of injury.

Exclusion Criteria:

* Patients with electrical burns, chemical burns, inhalation injury.
* Patients in overt shock (defined as serum lactate >2.5, or hypotension and altered mental status).
* Pregnant patients, psychiatrically unstable patients will be excluded.
* Patients with oropharyngeal defects and/or previously known diagnoses leading to high risk of aspiration, and/or precluding safe nasal-enteric access will be excluded.
* Patients will history of chronic nausea and/or vomiting, including those with a diagnosis of gastroparesis due to diabetes mellitus will be excluded.
* Patients with a Baux score of over 100 (age + TBSA), patients with declared palliative intent on admission, and patients for whom clinicians have high level of clinical concern based on clinical judgement will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kajal Mehta, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Nepal Cleft and Burn Center at Kirtipur Hospital, Ki̇̄rtipur, Bagmati, Nepal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 4 | 3 | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [32 to 61] | 50 [31 to 57.5] | 49 [30.5 to 59.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Nepal | 15 | 15 | 30
Total Body Surface Area (TBSA) with Burn Injury [Median (Inter-Quartile Range); unit: percentage of burned surface area] | 25 [21 to 32.5] | 30 [26 to 35.5] | 30 [22 to 35]

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Average Urine Output (UOP)
Description: Calculated by totaling all of the recorded urine output (adding up the columns labelled HR 1-2 UO, HR 3-4 UO, etc. until HR 23-24), then dividing by their weight in Kg (column labelled Admission weight) and dividing by 24 hours. The units of this measurement will be mL/kg/hr.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: ml/kg/hr
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
Number analyzed (Participants) | 15 | 15
ml/kg/hr | 0.7 [0.6 to 0.9] | 1 [0.7 to 1.2]

2. Primary Outcome: 24-hour Resuscitation Volume
Description: Calculated by totaling the total resuscitative fluids administered in first 24 hours of resuscitation, divided by admission weight and % TBSA of burn injury. (cc/kg/% TBSA of burn injury)
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: ml/kg/% of TBSA burned
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
Number analyzed (Participants) | 15 | 15
ml/kg/% of TBSA burned | 6.7 [5.4 to 9.9] | 4.1 [3.6 to 5.7]

3. Primary Outcome: Hours From Injury to Resuscitation
Description: Hours calculated from point of injury to starting of resuscitation.
Time Frame: Point measurement (Once at the start of resuscitation)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
Number analyzed (Participants) | 15 | 15
hours | 8.5 [4.3 to 12.5] | 13.5 [13 to 15.5]

4. Secondary Outcome: Number of Participants With GI Discomfort
Description: Any "check" for nausea, vomiting, distention, diarrhea
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
Number analyzed (Participants) | 15 | 15
Participants | 8 | 5

5. Secondary Outcome: Number of Participants Crossover to IV Due to GI Intolerance
Description: Number of participants crossover to standard of care (IV resuscitation) due to GI intolerance like nausea, vomitting
Time Frame: 24hours
Population: Not applicable to IV resuscitation arm as already on the standard of care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
Number analyzed (Participants) | 15 | 0
Participants | 9 | 0

6. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: Measured with any signs of Acute Kidney injury during first 72 hours of resuscitation according to KDIGO definition i.e., increase in serum creatinine by 0.3mg/dL or more within 48 hours or increase in serum creatinine to 1.5 times baseline or more within the last 7 days or urine output less than 0.5 mL/kg/h for 6 hours. AKI on admission was defined as a serum creatinine greater than 1.5 mg/dL with less than 0.5 mL/kg/h of urine output for the first hour. Urine output was measured every 2 hours for the first 24 hours and serum creatinine was measured on admission then 8,16,24,48 and 72 hours from the commencement of the resuscitation.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
Number analyzed (Participants) | 15 | 15
Participants
  On Admission | 4 | 2
  At 72 hours | 4 | 0
  Renal Failure within 72 hours | 1 | 0

7. Secondary Outcome: Participants Death Within 72 Hours of Resuscitation
Description: Secondary resuscitation outcome measured daily within study period i.e. 72 hours of resuscitation as participant death related or associated with the study. Monitored by data safety monitoring board and if proven to be associated with the study considered serious adverse event.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

8. Secondary Outcome: Discharge Outcome
Description: Outcome of hospital stay
Time Frame: Measured over complete course of hospitalization until discharge or death, assessed every 24 hours after enrollment in the study. Maximum timeframe 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
Number analyzed (Participants) | 15 | 15
Participants
  Discharged home | 6 | 5
  Left against medical advice | 3 | 6
  Death | 6 | 4

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Enteral-based Protocolized Resuscitation | Intravenous Fluid Protocolized Resuscitation
All-Cause Mortality (participants affected / at risk) | 6/15 | 4/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 8/15 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enteral-based Protocolized Resuscitation (N=15) | Intravenous Fluid Protocolized Resuscitation (N=15)
GI discomfort during resuscitation (Gastrointestinal disorders) | 8 | 5 — Check with any nausea, vomiting, distention, diarrhea during resuscitation period i.e. 24 hours

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT04732624/Prot_SAP_ICF_000.pdf